CLINICAL TRIAL: NCT06549400
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Once Daily Mexiletine PR in Patients With Myotonic Dystrophy Type 1 and Type 2 Who Have Completed the MEX-DM-302 Study (ATLAS Study)
Brief Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of Once Daily Mexiletine PR in Patients With Myotonic Dystrophy Type 1 and Type 2 Who Have Completed MEX-DM-302 Study.
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin Ltd. (Industry)
Collaborators: Lupin Atlantis Holdings S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEX-DM-303
Record Dates: First submitted 2024-05-09; First posted 2024-08-12 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Intervention Model Description: This is an open-label extension study intended to evaluate the continuous long-term (18 months) safety and efficacy of once daily mexiletine-prolonged release (mexiletine PR) for the symptomatic treatment of myotonia in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2) who have completed the parent study MEX-DM-302. The MEX-DM-302 is a multicenter, randomized, double-blind, parallel-group, placebocontrolled study intended to evaluate the safety and efficacy of mexiletine PR in patients with DM1 and DM2) for 6 months. At the completion of the final visit in Study MEX-DM-302 patients who continue to meet the eligibility criteria will be invited to rollover into this open-label study for an additional 18 months. All patients who elect to continue into this open-label study will receive active mexiletine PR (no placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mexiletine prolonged-release (PR) (Other): Mexiletine PR 167 mg (mexiletine HCl 200 mg) Mexiletine PR 333 mg (mexiletine HCl 400 mg) OR Mexiletine PR 500 mg (mexiletine HCl 600 mg)
  Interventions: Drug: Mexiletine granules for prolonged-release oral suspension

INTERVENTIONS:
Drug: Mexiletine granules for prolonged-release oral suspension — Mexiletine PR

SUMMARY:
This is an open-label extension study intended to evaluate the long-term safety and efficacy of mexiletine PR in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2) who have completed the parent study MEX-DM-302.

DETAILED DESCRIPTION:
At the completion of the final visit in Study MEX-DM-302 patients who continued to meet the eligibility criteria will be invited to rollover into this open-label study for an additional 18 months. All patients who elect to continue into this open-label study will receive active mexiletine (no placebo).

Mexiletine PR will be started as 167 mg once a day (QD) treatment regimen. The dose will be titrated up at Week 1 to 333 mg and at Week 2 to a maximum dose of 500 mg QD depending on tolerability. If unable to tolerate the escalated dose, the dose will be reduced by one dose step during the titration period of the study to a maximum tolerated dose. Study drug should be taken with food at approximately the same time of the day every day, preferably in the morning (See Section 7 for further details on reconstitution and dosing titration).

Safety assessments include patient- and physician-reported adverse events, standard clinical laboratory evaluations, physical examinations, and vital signs. In addition, ECG, Holter monitors, and echocardiogram assessments will be collected to assess cardiac safety during the study.

ELIGIBILITY:
Inclusion Criteria:

1. DM1 or DM2 diagnosis confirmed genetically;
2. Ability to comprehend and willingness to sign an informed consent (ICF) or ICF of the parent(s)/legal guardian and written assent from the patient (if patient < 18 years of age);
3. Ability to understand the study requirements including intention to stay in the study until the end-of-study visit at 26 weeks of treatment;
4. Male or non-pregnant female ≥16 years of age;
5. Body Mass Index (BMI) of 18.5 kg/m2 to 30 kg/m2, and weight ≥45 kg;
6. Female patients of childbearing potential must be using a highly effective form of birth control for the duration of the study and for at least 7 days after last dose of study drug;
7. No significant cardiac abnormalities as determined by a cardiologist's assessment;
8. Have sufficient finger flexor strength to grasp the handle of the dynamometer used to measure myotonia;
9. DM1 patients only - Muscular impairment rating scale (MIRS) score of 2, 3 or 4.

Exclusion Criteria:

1. Are pregnant or lactating;
2. Have any one of the following medical conditions: uncontrolled diabetes mellitus, cancer other than skin cancer less than five years previously (e.g., basal-cell carcinoma (BCC) and squamous-cell carcinoma (SCC) of skin allowed), multiple sclerosis, seizure disorders, or other serious medical illness;
3. Severe renal impairment (glomerular filtration rate (GFR) < 30 mL/min);
4. Medical conditions which could interfere with muscle function such as infections, trauma, fractures, or planned surgery;
5. Medical conditions that could affect hand functioning including but not limited to rheumatoid arthritis, Dupuytren's contracture, hand deformity, etc.;
6. Severe arthritis or medical condition (other thanDM1/DM2) that would significantly impact ambulation;
7. High incidence of falls or fall-associated fractures (>5 falls during the past 12 months);
8. Preexisting elevated liver function tests > 3 times the upper limit of normal (ULN) on Day 1 (alanine transaminase (ALT)/aspartate transaminase (AST), gamma-glutamyl transferase (GGT)) and/or any abnormal chemistry, hematology or urine lab considered clinically significant by investigator;
9. Serum potassium values < 3.5 mmol/L or > 5.0 mmol/L or serum magnesium values < 1.7 mg/dL. Electrolytic imbalance such as hypokalaemia, hyperkalaemia or hypomagnesaemia may increase the proarrhythmic effects of mexiletine. Electrolyte imbalances need to be corrected before administering mexiletine and will be monitored throughout treatment.
10. Intake of any anti-myotonic treatment within 4 weeks prior to baseline (Day 1) or 5 half-lives, whichever is longer such as metformin, such as propafenone, flecainide, lamotrigine, carbamazepine or any other channel-blocker/ anticonvulsive drugs;
11. Use of any concomitant medications that could increase the cardiac risk;
12. Known allergy to mexiletine or any local anesthetics;
13. Participation in another interventional clinical study during the last 3 months or 5 half-lives of the investigational medicinal product, whichever is longer (with the exception of participation in the previous MEX-DM-302 study);
14. Wheelchair-bound or bed-ridden;
15. Any cardiac safety associated condition including any of the following criteria detected by cardiac evaluations including 24-hr Holter monitor, echocardiogram and clinical evaluations:

    * PR interval ≥240 ms or QRS duration ≥120 ms on resting ECG
    * Personal history of 3rd degree or 2nd degree type 2 atrioventricular block or sinus node dysfunction with pauses ≥3 seconds, complete bundle branch block, bifascicular and trifascicular block or any heart block susceptible to evolve to complete heart block
    * Personal history of sustained atrial fibrillation, flutter or tachycardia (duration >30 seconds)
    * Personal history of non-sustained (ventricular triplets or more) or sustained ventricular tachycardia
    * Myocardial infarction (acute or past) or coronary artery stenosis >50%, presence of abnormal Q waves
    * New York Heart Association (NYHA) Class II to IV heart failure
    * Left ventricular systolic dysfunction with ejection fraction <50%
    * Sinus node dysfunction (including ECG sinus rate <50 beats per minute (BPM))
    * Co-administration of antiarrhythmics inducing torsades de pointes (class Ia: quinidine, procainamide, disopyramide, ajmaline; class Ic: encainide, flecainide, propafenone, moricizine; class III: amiodarone, sotalol, ibutilide, dofetilide, dronedarone, vernakalant)
    * Co-administration of other classes of antiarrhythmics (class Ib: lidocaine, phenytoin, tocainide; class II: propranolol, esmolol, timolol, metoprolol, atenolol, carvedilol, bisoprolol, nebivolol; class IV: verapamil, diltiazem)
    * Patients with implantable cardioverter defibrillators (ICDs) and pacemakers are excluded
    * Presence of symptomatic coronary artery disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2028-05-29 (Estimated); Study Completion 2028-07-06 (Estimated)

PRIMARY OUTCOMES:
To assess the long-term efficacy of once daily mexiletine PR for the symptomatic treatment of myotonia in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2) who have completed MEX-DM-302 study. | 78 weeks
  Handgrip relaxation time in DM1 patients by mean change in baseline of handgrip relaxation time (seconds) after maximal voluntary isometric contraction (MVIC)

SECONDARY OUTCOMES:
To assess the long-term safety of once daily mexiletine PR for the symptomatic treatment of myotonia in patients with myotonic dystrophy type 1 and type 2 (DM1 and DM2) who have completed the MEX-DM-302 study | 78 weeks
  Number and frequency of AEs/SAEs throughout the study while on treatment
Mean change in VAS | 78 weeks
  Score for muscle stiffness (myotonia severity) as self-reported by patients on a Visual Analog Scale (VAS)
Mean change in MBS scores | 78 weeks
  Mean change in Myotonia Behavior Scale (MBS) scores on a scale of 0 (no stiffness) to 5 (incapacitating stiffness)
Mean change in health-related quality of life | 78 weeks
  Mean change in health-related quality of life (measured by INQoL)
Mean change in DM1-Activ-c scale (DM1 patients only) | 78 weeks
  Mean change in measure of activity and social participation (measured by a Rasch-built scale with a 0-100 interval range)
Mean change in time to perform the 10-meter Walk Test | 78 weeks
  Mean change in time (seconds) to perform the 10-meter Walk Test (10mWT)
Mean change in handgrip relaxation time | 78 weeks
  Mean change in maximal voluntary isometric contraction (MVIC) and relaxation time by Video-recording of Hand Opening Time (VHOT) functional evaluation
Mean change in time to perform Timed-up and go (TUG) test | 78 weeks
  Mean change in time (seconds) to perform Timed-up and go (TUG) test
Mean change in health-related quality of life measured by EQ-5D | 78 weeks
  Mean change in health-related quality of life measured by EQ-5D (5-point scale)
Mean change in Myotonic Dystrophy Health Index (MDHI) score (DM1 patients) | 78 weeks
  Mean change in Myotonic Dystrophy Health Index (MDHI) score (DM1 patients) as measured by patient's perceived health
Mean change in Myotonic Dystrophy 2 Health Index (MD2HI) score (DM2 patients) | 78 weeks
  Mean change in Myotonic Dystrophy 2 Health Index (MDHI) score (DM2 patients) as measured by patient's perceived health
Assess the long-term safety of mexiletine PR by changes in ECG | 78 weeks
  Mean change in ECG (PR, QRS, and QTc intervals in units of milliseconds [ms]) from baseline
Assess the long-term safety of mexiletine PR by changes in ECG (HR) | 78 weeks
  Mean change in ECG (HR in units of beats per minute) from baseline
Assess the long-term safety of mexiletine PR by AEs | 78 weeks
  Incidence of treatment emergent adverse events (TEAEs), treatment-related TEAEs, serious AEs, and patient discontinuation rate
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (hematology measured in units of μL [microliters]) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by hematology parameters in units of μL: white blood cell (WBC) with differential (absolute count), red blood cells (RBC), platelet count, and red blood cell indicies.
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (hematology measured in units of % [percentage]) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by hematology parameters in units of %: white blood cell (WBC) and differential (percentage) and hematocrit.
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (hematology measured in g/dL [units of grams per deciliter]) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by hematology parameters in units of g/dL: hemoglobin.
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (chemistry measured in units of mmol/L) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by chemistry parameters in units of mmol/L: chloride, carbon dioxide, potassium, and sodium
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (chemistry measured in units of U/L) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by chemistry parameters in units of U/L: alkaline phosphatase, aspartate aminotransferase (AST), aspartate transaminase (ALT), gamma-glutamyl transferase (GGT), and creatine phosphokinase.
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (chemistry measured in units of g/dL) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by chemistry parameters in units of g/dL: albumin and total protein.
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (chemistry measured in units of mg/dL) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by chemistry parameters in units of mg/dL: blood urea nitrogen (BUN), calcium, creatinine (eGFR), glucose, total bilirubin, and magnesium.
Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations (urinalysis) from change in baseline | 78 weeks
  Assess the long-term safety of mexiletine PR by standard clinical laboratory evaluations as measured by urinalysis parameters (measured as normal or abnormal): appearance, specific gravity, pH, protein, glucose, ketones, blood, leukocyte esterase, nitrite, bilirubin, urobilinogen, and microscopic examination.
Assess the long-term safety of mexiletine PR by vital signs (pulse) | 78 weeks
  Assess the long-term safety of mexiletine PR by vital signs (pulse in units of bpm [beats per minute]) from change in baseline
Assess the long-term safety of mexiletine PR by vital signs (body temperature) | 78 weeks
  Assess the long-term safety of mexiletine PR by vital signs (body temperature in units of Fahrenheit or Celsius) from change in baseline
Assess the long-term safety of mexiletine PR by vital signs (blood pressure) | 78 weeks
  Assess the long-term safety of mexiletine PR by vital signs (blood pressure [diastolic and systolic] in units of mmHg [millimeters of mercury]) from change in baseline
Assess the long-term safety of mexiletine PR by vital signs (respiration) | 78 weeks
  Assess the long-term safety of mexiletine PR by vital signs (respiration in units of breaths per minute) from change in baseline
Assess the long-term safety of mexiletine PR by physical examinations | 78 weeks
  Assess the long-term safety of mexiletine PR by change in baseline from physical examinations (normal or abnormal) in the following regions and systems: general appearance, head and neck, heart, lung, abdomen, chest and back, upper extremities, lower extremities, neurological, and dermatological.

CONTACTS AND LOCATIONS:
Locations (6):
- Laboratory for Muscle Diseases and Neuropathies, Leuven, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- Ludug-Maximilians University, München, Germany
- Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Italy
- University Hospital of Madrid, Madrid, Spain
- University College Hospital, London, United Kingdom